CLINICAL TRIAL: NCT04533035
Title: Lower Limb Tissue Oxygenation Using Near-infrared Spectroscopy During Hallux Valgus Operation
Acronym: INVOHV
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Anna Govenius, Specialist in cardiothoracic surgery, MD, Kuopio University Hospital
Other Study IDs: 5101143
Record Dates: First submitted 2020-08-20; First posted 2020-08-31 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Lower Limb Ischemia
Keywords: NIRS Spectroscopy; Lower Limb; Ischemia; Adults
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort: 30 patients undergoing hallux valgus surgery

SUMMARY:
In acute lower limb ischemia the main goal of the treatment is to restore the blood before irreversible damage to the soft tissues of the limb. Delays in identifying acute lower limb ischemia may lead to limb loss or lead to the loss of the patient. Situations in which the patient is unable to express symptoms of the acute lower limb ischemia, such as during general anesthesia, in intensive care, or immediately after vascular surgery, are challenging for medical staff to identify. A reliable, easy-to-use and non-invasive monitoring method is not yet in every day use. The aim of this study is to demonstrate that Near InfraRed Spectroscopy (NIRS) monitoring is such a monitoring method.

Tourniquet induced ischemia is often used in hallux valgus surgery because it offers a bloodless view of the anatomical structures. In our study we will measure the soft tissue perfusion (rSO2) of the lower limbs during the whole operation. The sensors based on near-infrared spectroscopy will be located to the tibial surface and will record the normal state before the start of the tourniquet, during the tourniquet and also in the recovery phase.

The hypothesis is that rSO2 decreases linearly as a function of time from the beginning of the tourniquet induced ischemia and the recovery time depends on the duration of the tourniquet. In our study the patients will be operated under a spinal anesthesia. We also hypothesise that rSO2 increases due to the induction of the spinal anesthesia. Our goal is to define the percentual decline of rSO2 that is significant for lower limb ischemia and also its time response to induction of ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Patient understands the meaning of the study and related measures.
* Patient gives his or her written informed consent.
* A tourniquet is used.
* The procedure is performed under spinal anesthesia.
* Body mass index under 40.

Exclusion Criteria:

* Patient belongs to any of the following special groups: disabled people, minor, pregnant or breast feeding women, convicts, forensic psychiatric patients.
* Previous lower limb vascular surgery.
* Previous lower limb deep vein thrombosis.
* Previously performed tibial fasciotomies.
* Any another reason why the researcher considers that the patient is not suitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Operative hallux valgus patients in Kuopio University Hospital.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
The percentual decrease of the regional oxygen saturation in the lower limb 15 minutes after the tourniquet is applied. | 15 minutes from tourniquet application
  50% decrease from baseline NIRS value in 15 minutes

SECONDARY OUTCOMES:
The time that the regional oxygen saturation in the lower limb takes to recover after the tourniquet is released. | From the moment tourniquet is released to the point that NIRS value reaches it's baseline or patient is mobilised in the recovery room, whichever came first, assessed up to two hours.
  The time to NIRS value to reach baseline value after tourniquet is released
The percentual increase of the regional oxygen saturation in the lower limbs due to the induction of a spinal anesthesia. | 30 minutes from induction of spinal anesthesia
  10% increase in NIRS value after 30 minutes after spinal anesthesia induction

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo Mäkinen, docent, Study Director — Kuopio University Hospital; Anna H Govenius, MD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland